CLINICAL TRIAL: NCT06227754
Title: Randomized Controlled Trial of Optical Coherence Tomography Versus Angiography for Culprit Lesion Revascularization in Patients With Acute Myocardial Infarction
Brief Title: OCT Versus Angiography for Culprit Lesion Revascularization in Acute Myocardial Infarction PatiEnts
Acronym: FRAME-AMI3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Joon Hong, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRAMEAMI220716
Record Dates: First submitted 2023-12-31; First posted 2024-01-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: ST Elevation Myocardial Infarction; Myocardial Infarction
Keywords: ST-segment elevation MI; Optical coherence tomography; Intravascular imaging; Primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open-label, randomized controlled trial to compare clinical outcomes between optical coherence tomography (OCT)-guided versus angiography-guided PCI in AMI patients undergoing PCI.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography-guided PCI (Active Comparator): The PCI procedure in this group will be performed as standard procedure.
  Interventions: Procedure: Angiography-guided PCI group
- Optical coherence tomography-guided PCI (Experimental): Use of OCT will be allowed at any step of PCI (pre-PCI, during PCI and post-PCI), but OCT after stent implantation will be mandatory. In this group, the recommendations for selecting reference segment, selecting appropriate size of stent, and stent optimization are as follows. OPTIS imaging catheter (Abbott Vascular) will be used for the imaging arm according to MLD MAX algorithm.
  Interventions: Procedure: Optical coherence tomography-guided PCI group

INTERVENTIONS:
Procedure: Angiography-guided PCI group — The PCI procedure in this group will be performed as standard procedure. After deployment of stent, stent optimization will be done based on angiographic findings. The optimization guided by angiography should meet the criteria of angiographic residual diameter stenosis less than 10% by visual estimation and the absence of flow limiting dissection (≥Type C dissection). When angiographic under-expansion of the stent is suspected, adjunctive balloon dilatation will be strongly recommended.
  Arms: Angiography-guided PCI
Procedure: Optical coherence tomography-guided PCI group — [Stent Optimization]
  1. Stent Expansion:
     Visually assess residual angiographic diameter stenosis <10% "AND"
     ① In non-LM lesions: In-stent minimal lumen area (MSA) >80% of the average reference lumen area "OR" >4.5 mm2
     ② In LM lesion: MSA>7 mm2 for distal LM and >8 mm2 for proximal LM
  2. Stent Apposition:
     No major malapposition (defined as a distance from stent strut to adjacent intima ≥400 um and < 1mm length) of the stent over its entire length against the vessel wall
  3. Edge Dissection:
  No major edge dissection in the proximal or distal reference segments, defined as 5 mm from the edge of the stent, extended to media layer with potential to provoke flow disturbances (defined as >60° of the circumference of the vessel at site of dissection and/or >2 mm in length of dissection flap)
  Arms: Optical coherence tomography-guided PCI

SUMMARY:
The aim of the study is to compare clinical outcomes between optical coherence tomography-guided versus angiography-guided percutaneous coronary intervention (PCI) in patients with acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is a standard treatment for significantly stenotic lesion of coronary arteries, especially in the setting of acute myocardial infarction (AMI) where timely reperfusion is important. Traditionally, visual assessment by coronary angiography has been the main tool to identify coronary artery disease and guide revascularization. However, it is known that angiography alone is unable to adequately evaluate significance of stenotic lesion or optimization status of the stent, and that angiography suffers from high intra- and interobserver variability. Thus, methods for intracoronary imaging and/or physiology have been developed to aid these limitations.

During the PCI procedure, intravascular imaging devices such as intravascular ultrasound (IVUS) and optical coherence tomography (OCT) are useful tools for providing information on lesion characteristics and optimal stent implantation with regard to appropriate reference segment, stent expansion, stent apposition, and possible acute complications. Therefore, intravascular imaging guidance may improve clinical outcomes after complex PCI. However, although previous randomized controlled trial and registries showed significantly lower rates of major adverse clinical events following IVUS-guided PCI compared with angiography-guided PCI, the randomized controlled trials were limited with small sample size and dealt with very selected lesion subsets such as chronic total occlusion (CTO) or long lesions. Moreover, although some studies observed similar clinical outcomes between IVUS-guided PCI and OCT-guided PCI, it is uncertain whether OCT-guided PCI improves clinical outcomes compared with angiography-guided PCI.

Currently, randomized controlled trial to support beneficial impact of OCT-guided PCI, especially in patients with acute myocardial infarction (AMI) is lacking. One randomized clinical trial in 2016 with 240 non-ST-elevation myocardial infarction patients have reported higher postprocedural fractional flow reserve and similar incidence of major adverse cardiac events with the use of OCT compared to angiography alone, but this study mostly focused on immediate physiologic findings of OCT-guided PCI and only demonstrated clinical outcomes on short-term follow-up. Although the ILUMIEN IV trial evaluated efficacy of OCT-guided PCI among high risk patients including lesions were considered to be responsible for a recent myocardial infarction, there was no apparent difference in the target-vessel failure at 2 years. There is no randomized controlled trial that can provide information on its long-term clinical impact, and current clinical guidelines puts OCT on Class 2a recommendation as an alternative for IVUS, with the exception of ostial left main disease.

In this regard, randomized controlled trial comparing clinical outcome following PCI in patients with AMI where procedural optimization is performed under OCT-guidance or angiography alone would provide valuable evidence to enhance prognosis after treatment of AMI. Therefore, FRAME-AMI 3 trial has been designed to compare clinical outcomes after PCI for infarct-related artery using either OCT-guided or angiography-guided strategy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age
* Acute ST-segment elevation myocardial infarction (STEMI)

  *STEMI: ST-segment elevation ≥0.1 mV in ≥2 contiguous leads or documented newly developed left bundle-branch block1
* Primary percutaneous coronary intervention (PCI) in < 12 h after the onset of symptoms for STEMI patients
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

* Target lesions not amenable for PCI by operators' decision
* Ostial lesions located in left main vessel or right coronary artery (left main body or distal bifurcation lesions can be enrolled by operator's discretion)
* Creatinine clearance ≤30 ml/min/1.73 m2 and not on dialysis (chronic dialysis dependent patients are eligible for enrolment regardless of creatinine clearance)
* Cardiogenic shock (Killip class IV) at presentation
* Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, or Everolimus
* Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
* Pregnancy or breast feeding
* Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | 2 years after last patient enrollment
  a composite of cardiac death, target-vessel myocardial infarction, clinically-driven target-vessel repeat revascularization, definite or probable stent thrombosis

SECONDARY OUTCOMES:
All-cause death | 2 years after last patient enrollment
  All-cause death
Cardiac death | 2 years after last patient enrollment
  Cardiac death
Rate of any myocardial infarction | 2 years after last patient enrollment
  Any myocardial infarction, defined by Forth Universal definition of myocardial infarction
Rate of spontaneous myocardial infarction | 2 years after last patient enrollment
  Spontaneous myocardial infarction, defined by Forth Universal definition of myocardial infarction
Rate of procedure-related myocardial infarction | 2 years after last patient enrollment
  Procedure-related myocardial infarction, defined by ARC II definition
Rate of any revascularization | 2 years after last patient enrollment
  Any revascularization (clinically-driven or ischemia-driven)
Rate of target vessel revascularization | 2 years after last patient enrollment
  Target vessel revascularization
Rate of stent thrombosis | 2 years after last patient enrollment
  Definite or probable stent thrombosis, defined by ARC II definition
Total procedural time | at least 1 week after index procedure
  Total procedural time (primary PCI to end of the procedure including amount of staged procedure)
Total fluoroscopy time | at least 1 week after index procedure
  Total fluoroscopy time (primary PCI to end of the procedure including amount of staged procedure)
Total amount of contrast use | at least 1 week after index procedure
  Total amount of contrast use (primary PCI to end of the procedure including amount of staged procedure)
Incidence of contrast-induced nephropathy | at least 1 week after index procedure
  Incidence of contrast-induced nephropathy, defined as an increase in serum creatinine of ≥0.5mg/dL or ≥25% from baseline within 48-72 hours after contrast agent exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Young Joon Hong, MD, PhD, Principal Investigator — Chonnam National University; Joo-Yong Hahn, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (21):
- South Korea (21):
  - Dong-A University College of Medicine, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chonnam National University, Gwangju
  - Wonkwang University Hospital, Iksan
  - International St. Mary's Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Jeonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Kyung Hee University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - St. Carollo Hospital, Suncheon
  - Uijeongbu St Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
After publication of main paper, de-identified data will be shared upon reasonable requests after discussion by Executive Committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of main paper.
Access Criteria: Executive Committee will discuss to share the de-identified data upon reasonable requests.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT06227754/Prot_SAP_001.pdf